CLINICAL TRIAL: NCT07257705
Title: Evaluation of a Clinical Decision-Support App for Emergency Care in a Rural Ugandan Hospital: A Pilot Randomized Crossover Simulation Trial
Brief Title: Pilot Trial of a Clinical Decision-Support App for Managing Emergencies Among Clinicians in a Rural Ugandan Hospital
Acronym: OASES
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Michele Bombelli, Associate Professor, School of Medicine and Surgery, University of Milano-Bicocca, University of Milano Bicocca
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: UNIMIB-972-OASES; 2025-CONT-142-BiUniCrowd-OASES (Other Grant/Funding Number: University of Milano-Bicocca)
Record Dates: First submitted 2025-11-18; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Diarrhea Infectious; Seizures; Emergency Care; Clinical Decision Support Systems; Rural Health; Dyspnea
Keywords: OASES App; Clinical Decision Support Systems; Emergency Care; Simulation Trial
MeSH Terms: conditions — Dysentery; Seizures; Dyspnea | interventions — Organizations

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, stratified crossover simulation design. Each participant manages standardized emergency scenarios in two periods: one using the OASES App (intervention) and one using standard practice (control). The order of conditions is randomized with permuted blocks, stratified by cadre (nurse/nursing assistant vs. clinical officer) to ensure balance. A washout period of at least three days separates the two periods to minimize learning and carryover effects. Matched pairs of cases (A and B sets) are used to ensure comparable content between periods, and within each period the case order is randomized.
Who Masked: Outcomes Assessor
Masking Description: Independent outcome assessors who score participants' responses against gold-standard checklists are blinded to study allocation. They do not know whether the responses come from the OASES App-assisted or standard practice sessions. Participants, facilitators, and investigators are not masked due to the nature of the simulation design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OASES App-Assisted Emergency Care (Experimental): Participants will use the OASES tablet-based clinical decision-support system to manage simulated emergency cases of diarrhea, dyspnea, and seizures. The App incorporates the WHO Interagency Integrated Triage Tool (IITT) and evidence-based algorithms from WHO and Ugandan guidelines. It provides real-time guidance for triage, diagnosis, and treatment steps, while also collecting structured data. Before use, participants receive a short orientation to the App but no formal training.
  Interventions: Other: OASES App
- Standard Practice Emergency Care (No Intervention): Participants will manage the same simulated emergency cases of diarrhea, dyspnea, and seizures without the OASES App, using their usual knowledge, clinical experience, and available resources. Standard reference materials, including paper-based WHO Interagency Integrated Triage Tool (IITT) and Uganda Clinical Guidelines, are accessible. This arm reflects routine practice in the outpatient department of Dr. Ambrosoli Memorial Hospital.

INTERVENTIONS:
Other: OASES App — The OASES App is a tablet-based digital clinical decision-support system (CDSS) developed in 2025 by the University of Milano-Bicocca. The App digitizes validated WHO- and Uganda guideline-based triage and emergency care algorithms, including the Interagency Integrated Triage Tool (IITT) and condition-specific pathways for diarrhea, dyspnea, and seizures in both adults and children. It provides step-by-step guidance for frontline clinicians during emergency case management and simultaneously collects structured clinical data. The App is designed for offline use in rural hospitals with limited infrastructure. In this trial, participants receive a brief orientation but no formal training before using the App during simulation scenarios.
  Other Names: Organization for the Advancement and Support of Emergency Systems App; OASES Clinical Decision-Support App
  Arms: OASES App-Assisted Emergency Care

SUMMARY:
This study is testing a new mobile application called the OASES App, developed by the University of Milano-Bicocca. The App is designed to help frontline clinicians (nurses, clinical officers, and nursing assistants) provide faster and more accurate emergency care for patients with life-threatening conditions such as severe diarrhea, breathing difficulties, and seizures.

The OASES App guides clinicians step by step through internationally recognized emergency care guidelines, including triage, diagnosis, and treatment recommendations. It is intended to be used offline on a tablet, making it suitable for rural hospitals with limited resources.

This is a pilot study to understand whether the App improves the way clinicians manage simulated emergency cases compared to standard practice. About 16 clinicians at Dr. Ambrosoli Memorial Hospital, Kalongo, Uganda will take part in structured simulation exercises using realistic patient scenarios. Each participant will manage cases with and without the App, so that the two approaches can be compared.

The main goal is to evaluate whether the App helps clinicians follow evidence-based guidelines more consistently. Other goals include measuring accuracy of triage, diagnosis, and treatment decisions, as well as the time needed to complete cases and clinicians' perceptions of usability, trust, and feasibility.

No real patients will be involved in this study. All scenarios are simulations conducted in a safe, controlled environment. The results will help refine the App and inform the design of a larger study in the future.

DETAILED DESCRIPTION:
Emergency conditions such as severe diarrhea, dyspnea, and seizures remain major causes of morbidity and mortality in low- and middle-income countries. Despite the availability of World Health Organization (WHO) and national guidelines, adherence to evidence-based emergency practices is often suboptimal in rural health facilities. Common challenges include limited training, high workload, and lack of decision-support resources.

The Organization for the Advancement and Support of Emergency Systems (OASES) App was developed in 2025 by the University of Milano-Bicocca as part of a quality improvement collaboration with Dr. Ambrosoli Memorial Hospital, Kalongo, Uganda. The App digitizes validated emergency care algorithms derived from WHO frameworks and Ugandan clinical guidelines. It incorporates the Interagency Integrated Triage Tool (IITT) and provides structured pathways for the management of diarrhea, dyspnea, and seizures in both adults and children. Designed for offline use on Android tablets, the App offers step-by-step decision support for frontline clinicians while also collecting structured clinical data.

This pilot trial uses a randomized, stratified crossover simulation design to evaluate the effectiveness, usability, and feasibility of the OASES App before clinical deployment. Approximately 16 outpatient department (OPD) clinicians at Dr. Ambrosoli Memorial Hospital (including nurses, clinical officers, and nursing assistants) will participate. Each clinician will complete a total of 12 standardized emergency case scenarios, divided into two sessions: one using the OASES App and one using standard practice without the App. To minimize learning effects, sessions will be separated by at least a three-day washout period.

The case scenarios are adapted from WHO training materials (such as Basic Emergency Care and Emergency Triage Assessment and Treatment guidelines) and reflect typical emergency presentations seen in the hospital's OPD. Each participant will manage six scenarios per study arm (two diarrhea, two dyspnea, two seizures), designed in matched pairs for comparability. Scenarios are facilitated by trained researchers and scored against gold-standard checklists derived from WHO and Ugandan guidelines.

The primary objective of the study is to assess whether use of the OASES App improves clinicians' adherence to evidence-based management steps during simulated emergencies. Secondary objectives include assessing triage accuracy, diagnostic accuracy, appropriateness of disposition decisions, completeness of history-taking and physical examination (process quality), time required to complete cases, and clinician perceptions of usability, trust, and feasibility.

The trial involves no real patients; all activities are conducted in controlled, simulation-based environments. Risks to participants are minimal and mainly related to potential discomfort in being assessed. Benefits include the opportunity to practice emergency scenarios and become familiar with digital decision-support tools.

Data are collected electronically using Kobo Toolbox, with facilitator checklists, participant responses, and structured usability surveys. Responses are scored independently by two blinded assessors, with discrepancies resolved by consensus or third-party adjudication. Data will be analyzed using mixed-effects models appropriate for a crossover design.

Findings from this pilot trial will provide preliminary evidence on the effectiveness and acceptability of the OASES App among frontline clinicians in a rural African hospital. Results will inform refinement of the App, guide study procedures, and support the design of a larger powered trial. At a broader level, the study aims to contribute to the evidence base for digital health solutions to strengthen emergency and acute care in resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

* Nurses, clinical officers, or nursing assistants currently employed in the outpatient department (OPD) of Dr. Ambrosoli Memorial Hospital.
* Age ≥18 years.
* Willing and able to provide written informed consent.
* Available to participate in both simulation sessions.

Exclusion Criteria:

* Individuals unable or unwilling to participate in both scheduled simulation sessions.
* Individuals not currently employed in the OPD of Dr. Ambrosoli Memorial Hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Guideline-Adherent Management of Simulated Emergency Cases | Immediately after completion of each simulation scenario
  Proportion of pre-specified, evidence-based diagnostic and treatment actions (critical management steps) correctly performed by participants during simulated scenarios of diarrhea, dyspnea, and seizures. Performance will be scored against gold-standard checklists derived from WHO and Uganda clinical guidelines by two independent blinded assessors. The outcome is expressed as a proportion (0-1) of guideline-consistent critical management actions completed.

SECONDARY OUTCOMES:
Triage Accuracy | Immediately after completion of each simulation scenario
  Correct assignment of patients to Interagency Integrated Triage Tool (IITT) categories (Emergency/Red, Urgent/Yellow, Non-urgent/Green), compared to case-specific gold standards. Scoring performed by two blinded assessors.
Disposition Appropriateness | Immediately after completion of each simulation scenario
  Correctness of the decision to admit or discharge patients, compared to gold-standard expected dispositions derived from WHO and Ugandan guidelines. Scoring by two blinded assessors.
Diagnostic Accuracy | Immediately after completion of each simulation scenario
  Accuracy of working impression (initial stage) and final diagnosis (post-investigation stage), compared with case-specific gold-standard diagnoses. Scoring by two blinded assessors.
Guideline-Adherent Evaluation (Process Quality) | Immediately after completion of each simulation scenario
  Proportion of critical history and examination items elicited by clinicians during simulated cases, compared with case-specific lists from WHO guidelines. Scored by facilitators using structured checklists.
Time to Case Completion | Immediately after completion of each simulation scenario
  Duration in minutes required by participants to complete each simulated case, measured by facilitators during simulation sessions.
System Usability Scale (SUS) Score | Immediately after completion of the OASES App simulation session
  Usability of the OASES App measured by the validated 10-item System Usability Scale (SUS), completed by participants after simulation sessions involving the App. The scale ranges from 0 to 100, where higher scores indicate better usability.
Perceived Usefulness, Trust, Satisfaction, and Feasibility | Immediately after completion of the OASES App simulation session
  Clinicians' perceptions of the OASES App assessed through structured 5-point Likert-scale survey items (1 = strongly disagree to 5 = strongly agree), adapted from Technology Acceptance Model and related frameworks, and short qualitative debriefs.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Bombelli, MD, Principal Investigator — University of Milano Bicocca
Locations (1):
- Dr. Ambrosoli Memorial Hospital Kalongo, Kalongo, Agago District, Uganda

IPD SHARING:
Plan to Share IPD: No
This pilot study collects simulation-based performance data from a small number of clinicians. Because the dataset is small and involves individual-level performance in a professional setting, sharing could pose confidentiality risks despite de-identification. Aggregate results will be provided, but individual-level data will not be shared.

REFERENCES:
- See also: OASES Project Website — https://oasesresearch.org/